CLINICAL TRIAL: NCT03083405
Title: Evaluation of the Quality of Sleep, Endothelial Function, Cardiovascular Risk, Thyroid Function, a Function of Masticatory Muscles and Psycho-emotional State of Patients With Sleep Bruxism
Brief Title: Selected Disorders and Sleep Bruxism
Status: Enrolling by invitation | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Principal Investigator, Wroclaw Medical University
Other Study IDs: WMU1/2017
Record Dates: First submitted 2017-02-19; First posted 2017-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Bruxism; Hypertension; Thyroid Dysfunction; Mental Status Change; Sleep Apnea; Sleep Disorders; Cardiovascular Risk Factor; Cardiovascular Diseases; Temporomandibular Disorder
MeSH Terms: conditions — Sleep Bruxism; Hypertension; Sleep Apnea Syndromes; Sleep Wake Disorders; Cardiovascular Diseases; Temporomandibular Joint Disorders | interventions — Opipramol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Opipramol group: Patients diagnosed with SB and opipramol intervention.
  Interventions: Drug: Opipramol
- SB group: Patients diagnosed with SB and no drug intervention.
- Healthy controls: Patients without diagnosed SB.

INTERVENTIONS:
Drug: Opipramol — The study group will get a drug to decrease bruxism activity. Group will be evaluated using polysomnography included rhythmic masticatory muscle activity registration before and after intervention.
  Groups: Opipramol group

SUMMARY:
Sleep apnea is a common and serious health problem in the Polish population. According to epidemiological data problem concerns about 7% of the adult population. The most common sleep disorder is obstructive sleep apnea (OSA). The consequence of episodes of airway obstruction and sleep fragmentation is an inefficient sleep, pathological daytime sleepiness, falling asleep involuntarily, awakening with feelings of shortness of breath or throttling. The direct consequences of sleep apnea are hypoxia, increased heart rate and increased blood pressure. Frequent complications of OSA are hypertension, stroke, cardiac arrhythmia, coronary artery disease and pulmonary hypertension. An additional problem in patients with sleep apnea is an increased incidence of bruxism. Bruxism is a common problem; reports of prevalence range from 8-31% in the general population. The most common symptoms of bruxism include: hypersensitive teeth, tooth wear, damage to dental restorations (e.g. crowns and fillings), damage to periodontal and oral mucosa, masticatory muscle pain and headaches. The etiology of bruxism is multifactorial and not fully understood. It can be caused by biologic, psychologic and exogenous factors. Arousals during the apnea episodes are considered to be a major cause of sleep bruxism in OSA patients. The relationship between OSA and sleep bruxism is still not clearly defined. Further research is needed to help explain the relationship between these two phenomena, which will enable further therapy in patients with coexisting OSA and sleep bruxism (SB).

DETAILED DESCRIPTION:
1. Introduction Sleep apnea is a common and serious health problem in the Polish population. According to epidemiological data problem concerns about 7% of the adult population. The most common sleep disorder is obstructive sleep apnea (OBS). The essences of OBS are episodes of airway obstruction repeated many times during sleep. As a result the oxygen level in blood decreases. The result of increased muscle tension of upper respiratory tract and throat vibrations is a very loud snoring restoring breath. Episodes of apnea with arousals cause sleep fragmentation, shortage of deep sleep and rapid eye movement (REM). Such episodes occur repeatedly, several, or even dozens of times per hour of sleep. The consequence of episodes of airway obstruction and sleep fragmentation is an inefficient, lack of rest sleep, pathological daytime sleepiness, falling asleep involuntarily, awakening with feelings of shortness of breath or throttling. Fragmentation of sleep and repeated episodes of hypoxia result in deterioration of quality of life, chronic fatigue and an increased risk of communication accidents.

   The direct consequences of sleep apnea are hypoxia, awakening, increased heart rate and increased blood pressure. Frequent complications of obstructive sleep apnea (OSA) are hypertension, stroke, cardiac arrhythmia, coronary artery disease, pulmonary hypertension and heart failure. If left untreated, OSA contributes to the development of vascular endothelial dysfunction and increases the risk of premature death, especially in men under age of 50.

   An additional problem in patients with sleep apnea is an increased incidence of bruxism.

   Bruxism is a common problem; reports of prevalence range from 8-31% in the general population. The most common symptoms of bruxism include: hypersensitive teeth, tooth wear, damage to dental restorations (e.g. crowns and fillings), damage to periodontal and oral mucosa, masticatory muscle pain and headaches. Symptoms of bruxism may go unnoticed for a long time, which implies that patients often don't know about their condition. There are two different types of bruxism: Sleep Bruxism (SB) and Awake Bruxism (AB). Type SB consists of involuntary, episodic and rhythmic activity of masticatory muscles (Rhythmic Masticatory Muscle Activity / RMMA).

   The etiology of bruxism is multifactorial and not fully understood.It can be caused by biologic, psychologic and exogenous factors. Arousals during the apnea episodes are considered to be a major cause of sleep bruxism in OSA patients.

   The relationship between obstructive sleep apnea and sleep bruxism is still not clearly defined. Further research is needed to help explain the relationship between these two phenomena, which will enable further therapy in patients with coexisting OSA and SB.
2. Aim The aim of the study is evaluation of the quality of sleep, endothelial function, cardiovascular risk, thyroid function, a function of masticatory muscles, psycho-emotional status, genetic predispositions and drug effectiveness in patients with bruxism.
3. Methods The project will take place in the Sleep Laboratory at the Department of Internal Medicine, Occupational Diseases and Hypertension Medical University in Wroclaw. About 100 patients referred to the Department of Internal Medicine, Occupational Diseases and Hypertension and Clinical Oncology for suspected sleep apnea and bruxism will be included.

Patients from the Clinic of Prosthodontics operating at the Department of Prosthodontics, Medical University in Wroclaw and other dental institutions diagnosed using Diagnostic Criteria for Temporomandibular Disorders (DC / TMD) and Criteria of American Academy of Sleep Medicine International Classification of Sleep Disorders ICSD-3 evaluating bruxism will undergo polysomnography (PSG) with video recording.

Polysomnograms will be evaluated in a 30-second contributions, according to standard sleep criteria. PSG results will contain data on the latency of sleep, total sleep time (TST), sleep efficiency (%) and an evaluation of phases N1, N2, N3 and REM. Pathological respiratory events will be evaluated in accordance with the standards of the American Academy of Sleep. Apnea is defined as the absence of airflow through the respiratory tract by more than 10 seconds. The shallowness of breathing is defined as a decrease in respiratory amplitude by more than 30% for more than 10 seconds, with subsequent desaturation of more than 3% or subsequent awakening.

Then, to evaluate the function of vascular endothelium in patients expansion of the brachial artery using ultrasonography Aloka Prosound Alpha 6, using the guidelines of the international working group studying reactivity of the brachial artery will be explored. Ultrasound of the heart, Electrocardiography Holter and Ambulatory blood pressure monitoring (ABPM) will be performed in each patient. In addition, researchers will execute surveys: Epworth Scale, Athens Scale, STOP-Bang Scale, Berlin questionnaire, the severity level of fatigue / tiredness scale, a questionnaire assessing quality of life, the scale of perceived stress - questionnaire PSS 10 and questionnaires Oral Behavior Checklist (OBC) and Pittsburgh Sleep Quality index (PSQI). Headache episodes will be assessed using Headache Impact Test - 6 (HIT-6) and HUNT questionnaires.

Each patient will be performed laboratory blood tests to determine levels of FT3, FT4 and TSH in order to evaluate the relationship between RMMA and thyroid disease and genetical tests. At the same time the relationship between bruxism, psycho-emotional state and sleep quality will be evaluated through questionnaires PSS10, OBC and PSQI.

Masticatory muscle activity during the study will be assessed on the basis of the record coming from electromyography electrodes placed on the beard and symmetrically around the masseter muscle attachments. The results will then be analyzed for the incidence RMMA directly related to episodes of bruxism and their relation to episodes of sleep apnea, changes in blood pressure and heart rate to determine the prevalence of cause-effect relationships.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed sleep bruxism
* full dentition
* single tooth loss
* age between 18 and 70

Exclusion Criteria:

* age under 18
* age over 70
* terminal general diseases
* severe mental disorders
* edentulism
* taking drugs that could falsify polysomnography
* confirmed alcoholism
* drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the Clinic of Prosthodontics operating at the Department of Prosthodontics, Medical University in Wroclaw and other dental institutions diagnosed with sleep bruxism using Diagnostic Criteria for temporomandibular Disorders (DC / TMD). Patients referred to the Department of Internal Medicine, Occupational Diseases and Hypertension and Clinical Oncology for suspected sleep apnea and bruxism. Healthy controls.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between bruxism and quality of sleep assessed by polysomnography. | 01.03.2017 - 01.03.2018
  Polysomnograms will be evaluated in a 30-second contributions, according to standard sleep criteria. PSG results will contain data on the latency of sleep, total sleep time (TST), sleep efficiency (%) and an evaluation of phases N1, N2, N3 and REM.

SECONDARY OUTCOMES:
Relationship between bruxism and quality of sleep assessed by Epworth scale. | 01.03.2017 - 01.03.2018
  Each participant will fill in Epworth scale.
Relationship between bruxism and quality of sleep assessed by Athens scale. | 01.03.2017 - 01.03.2018
  Each participant will fill in Athens scale.
Relationship between bruxism and quality of sleep assessed by STOP-bang questionnaire. | 01.03.2017 - 01.03.2018
  Each participant will fill in STOP-bang questionnaire.
Relationship between bruxism and quality of sleep assessed by Pittsburgh Sleep Quality Index. | 01.03.2017 - 01.03.2018
  Each participant will fill in Pittsburgh Sleep Quality Index.
Relationship between bruxism and sleep apnea assessed by polysomnography and genetical tests. | 01.03.2017 - 01.03.2018
  Each participant will fill undergo polysomnography and genetical blood tests.
Relationship between bruxism and sleep apnea assessed by Berlin questionaire. | 01.03.2017 - 01.03.2018
  Each participant will fill in Berlin questionaire.
Relationship between bruxism and cardiovascular risk assessed by ABPM. | 01.03.2017 - 01.03.2018
  Cardiovascular risk will be assessed in each participant using ABPM.
Relationship between bruxism and cardiovascular risk assessed by ECG Holter. | 01.03.2017 - 01.03.2018
  Cardiovascular risk will be assessed in each participant using ECG Holter.
Relationship between bruxism and cardiovascular risk assessed by heart ultrasonography. | 01.03.2017 - 01.03.2018
  Cardiovascular risk will be assessed in each participant using heart ultrasonography.
Relationship between bruxism and the function of vascular endothelium assessed by expansion of the brachial artery using ultrasonography. | 01.03.2017 - 01.03.2018
  Expansion of the brachial artery will be evaluated using ultrasonography Aloka Prosound Alpha 6.
Relationship between bruxism and thyroid function assessed by clinical tests of blood. | 01.03.2017 - 01.03.2018
  Blood test determining levels of FT3, FT4, TSH and Anti-TPO will be conducted for each participant to evaluate the function of thyroid.
Relationship between bruxism and masticatory muscle activity assessed by electromyography. | 01.03.2017 - 01.03.2018
  Masticatory muscle activity during the study will be assessed on the basis of the record coming from EMG electrodes placed on the beard and symmetrically around the masseter muscle attachments.
Relationship between bruxism, quality of life and mental status assessed by the scale of perceived stress - questionnaire PSS 10. | 01.03.2017 - 01.03.2018
  Each participant will fill in the scale of perceived stress - questionnaire PSS 10.
Relationship between bruxism, quality of life and mental status assessed by the questionnaire assessing quality of life. | 01.03.2017 - 01.03.2018
  Each participant will fill in a questionnaire assessing quality of life.
Relationship between bruxism quality of life and mental status assessed by the severity level of fatigue scale. | 01.03.2017 - 01.03.2018
  Each participant will fill in severity level of fatigue scale.
Relationship between bruxism quality of life and mental status assessed by the severity level of tiredness scale. | 01.03.2017 - 01.03.2018
  Each participant will fill in severity level of tiredness scale.
Relationship between bruxism and mental status assessed by Beck Depression Inventory | 01.03.2017 - 01.03.2018
  Each participant will fill in Beck Depression Inventory.
Relationship between bruxism and temporomandibular disorders (TMD). | 01.03.2017 - 01.03.2018
  Each participant will fill in TMD pain screener, Oral Behavior Checklist. All of the participants will also undergo diagnostics in accordance to DC/TMD.
Relationship between bruxism and headaches assessed by Headache Impact Test - 6 (HIT-6). | 01.03.2017 - 01.03.2018
  Each participant will fill in HIT-6 questionnaire.
Relationship between bruxism and headaches assessed by HUNT questionnaire. | 01.03.2017 - 01.03.2018
  Each participant will fill in HUNT questionnaire.
Effect of treatment with opipramol on bruxism episodes. | 01.03.2017 - 01.03.2018
  Opipramol treatment will be implemented in patients with bruxism.
Is bruxism genetically determined? | 01.03.2017 - 01.03.2018
  Each patient will undergo genetical blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Martynowicz, M.D., Ph.D., Principal Investigator — Wroclaw Medical University; Mieszko Wieckiewicz, D.M.D., Ph.D., Study Chair — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wieczorek T, Wieckiewicz M, Smardz J, Wojakowska A, Michalek-Zrabkowska M, Mazur G, Martynowicz H. Sleep structure in sleep bruxism: A polysomnographic study including bruxism activity phenotypes across sleep stages. J Sleep Res. 2020 Dec;29(6):e13028. doi: 10.1111/jsr.13028. Epub 2020 Mar 11. PMID 32160378
- [Derived] Smardz J, Martynowicz H, Wojakowska A, Michalek-Zrabkowska M, Mazur G, Wieczorek T, Wieckiewicz M. The meaning of the masticatory muscle tonic-type electromyographic pathway correlated with sleep bruxism and sleep-related breathing disorders - A polysomnographic study. Sleep Med. 2020 Apr;68:131-137. doi: 10.1016/j.sleep.2019.08.025. Epub 2019 Oct 2. PMID 32035303
- [Derived] Martynowicz H, Smardz J, Michalek-Zrabkowska M, Gac P, Poreba R, Wojakowska A, Mazur G, Wieckiewicz M. Evaluation of Relationship Between Sleep Bruxism and Headache Impact Test-6 (HIT-6) Scores: A Polysomnographic Study. Front Neurol. 2019 May 14;10:487. doi: 10.3389/fneur.2019.00487. eCollection 2019. PMID 31139138
- [Derived] Smardz J, Martynowicz H, Michalek-Zrabkowska M, Wojakowska A, Mazur G, Winocur E, Wieckiewicz M. Sleep Bruxism and Occurrence of Temporomandibular Disorders-Related Pain: A Polysomnographic Study. Front Neurol. 2019 Mar 11;10:168. doi: 10.3389/fneur.2019.00168. eCollection 2019. PMID 30915015